CLINICAL TRIAL: NCT02464774
Title: Impact of Breast-Conserving Therapy (BCT) on Recurrence in Patients With Triple-Negative Breast Cancer (TNBC) Compared With Mastectomy
Brief Title: Breast-Conserving Therapy in Patients With Triple-Negative Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaoming Xie (Other)
Responsible Party: Sponsor-Investigator, Xiaoming Xie, Chief, Department of Breast Surgical Oncology,Sun Yat-sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-FXY-093
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Triple-Negative Breast Cancer; Breast-Conserving Therapy; Mastectomy; Recurrence
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Recurrence | interventions — Mastectomy, Segmental; Mastectomy; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breast-Conserving Therapy (Experimental): 1. Patients undergo lumpectomy with surgical axillary staging with all lesions resected to negative margins.
  2. Within 4-8 weeks after surgery, patients receive adjuvant chemotherapy as follows:
     TC for stage I: Docetaxel 75 mg/m + Cyclophosphamide 600 mg/m, cycled every 21 days for 4 cycles.
     TAC for stage II: Docetaxel 75 mg/m + Doxorubicin 50 mg/m + Cyclophosphamide 500 mg/m, cycled every 21 days for 6 cycles.
  3. Within 4-8 weeks after completion of chemotherapy, patients undergo radiation therapy as follows:
  N0: Radiation therapy to whole breast (+boost to tumor bed). N1: Radiation therapy to whole breast (+boost to tumor bed), infraclavicular region, and supraclavicular area with or without radiation therapy to internal mammary nodes.
  Interventions: Procedure: Breast-Conserving Therapy; Drug: Adjuvant Chemotherapy; Radiation: Radiation Therapy
- Mastectomy (Active Comparator): 1. Patients undergo mastectomy (MT) with surgical axillary staging.
  2. Within 4-8 weeks after surgery, patients receive adjuvant chemotherapy as follows:
  TC for stage I: Docetaxel 75 mg/m + Cyclophosphamide 600 mg/m, cycled every 21 days for 4 cycles.
  TAC for stage II: Docetaxel 75 mg/m + Doxorubicin 50 mg/m + Cyclophosphamide 500 mg/m, cycled every 21 days for 6 cycles.
  Interventions: Procedure: Mastectomy; Drug: Adjuvant Chemotherapy

INTERVENTIONS:
Procedure: Breast-Conserving Therapy — Patients undergo lumpectomy with surgical axillary staging with all lesions resected to negative margins.
  Arms: Breast-Conserving Therapy
Procedure: Mastectomy — Patients undergo mastectomy with surgical axillary staging with all lesions resected to negative margins.
  Arms: Mastectomy
Drug: Adjuvant Chemotherapy — Patients with stage I and II receive adjuvant chemotherapy using TC and TAC regimen respectively.
Radiation: Radiation Therapy — N0: Radiation therapy to whole breast (+boost to tumor bed) or consideration of partial breast irradiation in selected patients; (2) N1: Radiation therapy to whole breast (+boost to tumor bed), infraclavicular region, and supraclavicular area with or without radiation therapy to internal mammary nodes.
  Arms: Breast-Conserving Therapy

SUMMARY:
RATIONALE: Triple-negative breast cancer (TNBC) is an aggressive subtype shown to have a high risk of locoregional recurrence (LRR) and distant metastasis (DM). The equivalent impact of breast-conserving therapy (BCT) and mastectomy on disease-free survival in patients with early breast cancer has been established by a number of large randomized controlled trials and meta-analysis. However, ongoing dispute exists on whether TNBC is a good candidate for BCT.

PURPOSE: This prospective, randomized, open, single-center Phase III clinical study is conducted to compare efficacy and safety of breast-conserving therapy and mastectomy in treating Chinese patients with early TNBC.

DETAILED DESCRIPTION:
STUDY POPULATION:

Operable patients with T1-2N0-1M0 triple-negative breast cancer

OBJECTIVES:

Primary To assess the impact of breast-conserving therapy on disease-free survival compared with mastectomy in patients with T1-2N0-1M0 triple-negative breast cancer.

Secondary To assess the impact of breast-conserving therapy on locoregional recurrence-free survival (LRRFS) and distant metastasis-free survival (DMFS) compared with mastectomy in patients with T1-2N0-1M0 triple-negative breast cancer.

OUTLINE:

This is a prospective, randomized, open, single-center Phase III clinical study.

Patients undergo either lumpectomy or mastectomy with surgical axillary staging with all lesions resected to negative margins based on the results of randomization generated by computer.

Patients with stage I and II receive adjuvant chemotherapy using TC and TAC regimen respectively.

Since all tumors are smaller than 5cm and metastatic lymph nodes are less than 4, patients undergoing mastectomy do not receive radiation therapy. On the hand, within 4-8 weeks after completion of chemotherapy, patients undergoing breast-conserving surgery receive radiation therapy as follows: (1) N0: Radiation therapy to whole breast (+boost to tumor bed) or consideration of partial breast irradiation in selected patients; (2) N1: Radiation therapy to whole breast (+boost to tumor bed), infraclavicular region, and supraclavicular area with or without radiation therapy to internal mammary nodes.

After completion of study treatment, patients are followed up every 3 months for 2 years and then 6 months for years 3-5.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 - 65 years old;
2. Staging of Cancer: cT1-2N0-1M0;
3. Histological confirmed with unilateral invasive carcinoma (all pathological types are applicable);
4. Definite reports on ER/PR/Her2 receptor showing all ER/PR/Her2 negative (specific definitions: immunohistochemical detection of ER <10% tumor cells is defined as ER negative, PR <10% positive tumor cells is defined as PR-negative, Her2 is 0~1+ or 2+ but determined negative via FISH or CISH detected (no amplification) is defined as Her2 negative);
5. Newly diagnosed conditions allowing direct surgery without any absolute contraindication for surgery;
6. ECOG performance score is 0 or 1;
7. No mass or microscopic tumor residue after surgery resection;
8. Informed consent form signed.
9. Willing to return to enrolling institution for follow-up during the Active Monitoring Phase (the active treatment and observation portions) of the study.

Exclusion Criteria:

1. Bilateral breast cancer;
2. Clinical or radiographic evidence of metastatic disease;
3. Widespread disease that cannot be incorporated by local excision through a single incision that achieves negative margins with a satisfactory cosmetic result;
4. Diffuse suspicious or malignant-appearing microcalcifications;
5. Positive pathologic margin;
6. Any of ER, PR or Her2 is positive;
7. Previous neoadjuvant therapy, including chemotherapy, radiotherapy and hormone therapy;
8. Prior history of breast cancer or any other malignant disease (except for basal cell carcinoma and cervical carcinoma in situ);
9. Severe systemic disease and/or uncontrollable infection, unable to be enrolled in this study;
10. Known allergic to taxane and anthracycline agents;
11. Pregnant and breast-feeding women;
12. With mental illness and cognitive impairment, unable to understand trial protocol and side effects and complete trial protocol and follow-ups;
13. Without personal freedom and independent civil capacity.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2015-07; Primary Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival(DFS) | Up to 5 years post-treatment
  DFS is defined as time (measured in months) from initial local-regional surgical treatment until first recurrence (local or distant) or last follow-up.

SECONDARY OUTCOMES:
Locoregional recurrence-free survival(LRRFS) | Up to 5 years post-treatment
  LRR refers to any progression in the breast/chest wall and/or regional lymph nodes.
Distant metastasis (DM) | Up to 5 years post-treatment
  DM is determined by clinical and radiographic means and/or histologically proven larger than 0.2mm.